CLINICAL TRIAL: NCT02968589
Title: @ctiveHip: Tele-rehabilitation System for Hip Fracture Patients
Brief Title: @ctiveHip Tele-rehabilitation System
Acronym: @ctiveHip
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Granada (Other)
Collaborators: Complejo Hospitalario Universitario de Granada (Other); Andalusian Initiative for Advanced Therapies - Fundación Pública Andaluza Progreso y Salud (Other)
Responsible Party: Principal Investigator, Patrocinio Ariza Vega, PhD, Universidad de Granada
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: University Hospital of Granada
Record Dates: First submitted 2016-11-13; First posted 2016-11-18 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Hip Fractures
Keywords: Tele-rehabilitation; Function; Quality of life; Exercise; Occupational Therapy; Physiotherapy; Caregiver burden
MeSH Terms: conditions — Hip Fractures; Motor Activity; Caregiver Burden

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- @ctiveHip intervention (Experimental): A training session for caregivers of patients with hip fracture on patient management.
  The @ctiveHip tele-rehabilitation system. This system includes a 3-months occupational therapy and exercise-based program, recommendations for patients and their caregivers and the option of chats and videoconferences.
  The program consists of 5 sessions/week of 50-60 minutes that patients will do at home. Each session includes videos with the prescribed activities and exercises that the patients will find in the private site of www.activehip.es.
  Interventions: Behavioral: Training
- Other training (Active Comparator): A training session for caregivers of patients with hip fracture on patient management.
  The usual care for hip fracture patients at hospital discharge. In addition, patients and their families will receive a triptych with information on recommendations and exercises to do at home.
  Interventions: Behavioral: Training

INTERVENTIONS:
Behavioral: Training

SUMMARY:
The purpose of this study is to determine if the @ctivehip tele-rehabilitation system improves the functional level and quality of life of hip fracture patients and reduce the caregiver burden.

DETAILED DESCRIPTION:
Background: The best option for rehabilitation after a hip fracture is still unclear. The home rehabilitation is one of the options and the use of tele-rehabilitation programs at home could be the option for some patients in the future. The main objective of this study is to improve the functional level and quality of life of hip fracture patients and reduce the caregiver burden using the @ctivehip tele-rehabilitation system.

Methods: This project will include hip fracture patients who met the following inclusion criteria: having a high pre-fracture functional level, not having severe cognitive impairment, absence of terminal disease, absence of post-surgery complications, going to live to their home or a relative home at hospital discharge, and signing an informed consent. The criteria to be part of this experimental group will be: having internet at home and a main caregiver with the ability to use the internet (@ctiveHip system). Patients without the internet at home will be part of the no intervention group, and they will receive the usual care, in addition to a triptych with information on recommendations and exercises to do at home. Caregivers of patients of both groups will receive a training session on patient management. Patients will be assessed at 4-weeks and 12 weeks after beginning to use the @ctiveHip system. The primary outcome will be the Functional level, measured by the Functional Independence Measure. The secondary outcomes: quality of life (Euro-qol), physical function (Timed Up and Go, Short Physical Performance Battery, International Fitness Scale), emotional status ( The Hospital Anxiety and Depression Scale ), health status (American Society of Anesthesiologists Score), cognitive status (Mini-mental Test ), fear of falling (Short Falls efficacy scale), pain (visual analogue scale), and caregiver burden of care (Zarit Burden Interview).

Discussion: This study has been designed to provide a tele-rehabilitation system which includes a rehabilitation protocol created by a multidisciplinary team of surgeons, occupational therapist, physiotherapist, and sport scientist, to improve the functional level of patients after hip fracture surgery. The @ctiveHip system could be a new low cost treatment option for some hip fracture patients.

ELIGIBILITY:
Inclusion Criteria:

Patients who had hip fracture surgery

Having a high pre-fracture functional level

Having Internet at home

Hospital discharge to their homes or a relative home.

A main caregiver who has the ability to use the internet (@ctivehip system)

Have signed an informed consent

Exclusion Criteria:

Presence of severe cognitive impairment

Presence of terminal disease

Presence of post-surgery complications

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Functional Level | Participants will be followed over 12 weeks
  The primary outcome will be assessed with the Functional Independence Measure, which is one of the most widely used instruments to measure Functional Level of hip fracture patients.

SECONDARY OUTCOMES:
Quality of life | 12 weeks
  The secondary outcome will be assessed with the EuroQoL Quality of Life Questionnaire which is one of the most widely used instruments to measure quality of life of hip fracture patients.
Mobility | 12 weeks
  Timed Up and Go test will be used to measure physical function.
Physical Function | 12 weeks
  Short Physical Performance Battery will be used to measure physical function.
Fitness | 12 weeks
  International Fitness Scale will be used to evaluate perceived patient´s overall fitness, cardio-respiratory fitness, muscular fitness, speed-agility and flexibility.
Emotional status | 12 weeks
  The Hospital Anxiety and Depression Scale will be used to evaluate the emotional status
Health Status | 12 weeks
  Health Status will be assessed using the American Society of Anesthesiologists Score
Cognitive status | 12 weeks
  Mini-mental Test will be used to measure the cognitive status of hip fracture patients.
Fear of falling | 12 weeks
  Short Falls Efficacy Scale will be used to assess fear of falling
Pain | 12 weeks
  The pain will be assessed using the Visual Analogue Scale
Caregiver burden | 12 weeks
  Zarit Burden Interview will be used to evaluate the caregiver burden of care

CONTACTS AND LOCATIONS:
Locations (1):
- Complejo Hospitalario Universitario de Granada, Granada, Spain

REFERENCES:
- [Derived] Prieto-Moreno R, Molina-Garcia P, Ortiz-Pina M, Mora-Traverso M, Estevez-Lopez F, Martin-Matillas M, Ariza-Vega P. Association of the @ctivehip tele-rehabilitation with the fear of falling of older adults with hip fracture and their family caregivers: Secondary analysis of a non-randomised controlled trial. J Telemed Telecare. 2025 Sep;31(8):1152-1161. doi: 10.1177/1357633X241257972. Epub 2024 Jun 5. PMID 38836335
- [Derived] Mora-Traverso M, Prieto-Moreno R, Molina-Garcia P, Salas-Farina Z, Martin-Martin L, Martin-Matillas M, Ariza-Vega P. Effects of the @ctivehip telerehabilitation program on the quality of life, psychological factors and fitness level of patients with hip fracture. J Telemed Telecare. 2024 Apr;30(3):549-558. doi: 10.1177/1357633X211073256. Epub 2022 Jan 21. PMID 35060784
- [Derived] Ariza-Vega P, Prieto-Moreno R, Castillo-Perez H, Martinez-Ruiz V, Romero-Ayuso D, Ashe MC. Family Caregivers' Experiences with Tele-Rehabilitation for Older Adults with Hip Fracture. J Clin Med. 2021 Dec 13;10(24):5850. doi: 10.3390/jcm10245850. PMID 34945145
- [Derived] Ortiz-Pina M, Molina-Garcia P, Femia P, Ashe MC, Martin-Martin L, Salazar-Gravan S, Salas-Farina Z, Prieto-Moreno R, Castellote-Caballero Y, Estevez-Lopez F, Ariza-Vega P. Effects of Tele-Rehabilitation Compared with Home-Based in-Person Rehabilitation for Older Adult's Function after Hip Fracture. Int J Environ Res Public Health. 2021 May 20;18(10):5493. doi: 10.3390/ijerph18105493. PMID 34065523
- [Derived] Ortiz-Pina M, Salas-Farina Z, Mora-Traverso M, Martin-Martin L, Galiano-Castillo N, Garcia-Montes I, Cantarero-Villanueva I, Fernandez-Lao C, Arroyo-Morales M, Mesa-Ruiz A, Castellote-Caballero Y, Salazar-Gravan S, Kronborg L, Martin-Matillas M, Ariza-Vega P. A home-based tele-rehabilitation protocol for patients with hip fracture called @ctivehip. Res Nurs Health. 2019 Feb;42(1):29-38. doi: 10.1002/nur.21922. Epub 2018 Nov 16. PMID 30444530